CLINICAL TRIAL: NCT01016925
Title: Bacterial Colonization After Tunneling in Femoral Perineural Catheters
Acronym: Tunnelized KT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2008/065/HP
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Bacterial Colonization
Keywords: femoral perineural catheter; tunnelization; complication; colonization; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control (No Intervention)
- femoral tunnelized perineural catheter (Experimental)
  Interventions: Procedure: tunnelized perineural catheter

INTERVENTIONS:
Procedure: tunnelized perineural catheter — the catheter will be tunneled 2-3 cm subcutaneously.
  Arms: femoral tunnelized perineural catheter

SUMMARY:
Background: Bacterial colonization of peripheral nerve catheters is frequent, although infection is relatively rare. With central venous catheters, the tunneling of catheter into the subcutaneous tissue significantly decreases catheter colonization and catheter-related sepsis.

Purpose: The aim of this study is to evaluate the incidence of bacterial colonization in adult patients with femoral tunnelized perineural nerve catheters.

Methods: A total of 338 patients with femoral catheter will be included in the study. The patients will be randomized to be included in the control group (without tunnelling) or in the group with catheter tunneled 2-3 cm subcutaneously. After removal, catheter will be analyzed for colonization (primary outcome). Quantitative culture will be used as described by Brun-Buisson for intravascular catheters. The site of insertion will be monitored daily for any signs of infection (secondary outcome).

Perspective: To show the incidence of femoral perineural catheter colonization is low with subcutaneous tunneling

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo scheduled orthopaedic surgery performed with a femoral perineural catheter

Exclusion Criteria:

* Age under 18 years
* Local nerve pathology
* Refusal to regional anaesthesia
* Major psychological disorder
* Major cardiac conduction disease
* Infection at the puncture site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
incidence of femoral perineural catheter colonization | between 24 hours and 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France